CLINICAL TRIAL: NCT07148011
Title: Radicle Revive™ CSP: A Randomized, Double-Blind, Placebo-Controlled, Trial Evaluating Plant-Based Health and Wellness Products on Perimenopausal Women's Self-Reported Health Issues and Outcomes
Brief Title: Radicle Revive™ CSP: A Trial Evaluating Plant-Based Health and Wellness Products on Perimenopausal Women's Self-Reported Health Issues and Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX_C_2507_SP
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-08

CONDITIONS: Perimenopause

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on their age and health outcome score during enrollment then randomized to one of the study arms. Each participant will have an equal chance of being assigned to each study arm.
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants' assigned study products. Participants are blinded to the study product they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Control (Placebo Comparator): Revive Product Form - Control
  Interventions: Dietary Supplement: Revive Product Form - Placebo Control
- Active Product (Experimental): Revive Product Form - Active
  Interventions: Dietary Supplement: Revive Product Form - Active

INTERVENTIONS:
Dietary Supplement: Revive Product Form - Placebo Control — Participants will use their Revive Product Form - Placebo Control as directed for a period of 12 weeks.
  Arms: Placebo Control
Dietary Supplement: Revive Product Form - Active — Participants will use their Revive Product Form - Active as directed for a period of 12 weeks.
  Arms: Active Product

SUMMARY:
A randomized, double-blind, placebo-controlled, trial evaluating plant-based health and wellness products on perimenopausal women's self-reported health issues and outcomes

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study conducted with adult participants, residing in the United States.

Eligible participants (1) are female, (2) are perimenopausal, (3) have the opportunity for meaningful improvement (at least 30%) in their primary health outcome, and (4) express acceptance in taking study products and not knowing the formulation identities until the end of the study.

Participants that report a known cardiac dysfunction, liver or kidney disease may be excluded. Participants that report a known contraindication or with well-established, significant safety concerns due to illness will be excluded. Heavy drinkers and women who are pregnant, trying to become pregnant, or breastfeeding will be excluded. Participants that report taking medications with a known contraindication or with well-established, significant safety concerns will be excluded.

Self-reported data are collected electronically from eligible participants for 13 weeks. Participant reports of health indicators will be collected at baseline, throughout the active period of study product use, and in a final survey. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
Inclusion Criteria:

* Adults, aged 37 - 55 years at the time of electronic consent, inclusive of all ethnicities, races, and gender identities
* Assigned sex at birth is female
* Resides in the United States
* Identifies menstrual status as perimenopausal
* Has the opportunity for at least 30% improvement in their primary health outcome
* Expresses a willingness to take a study product and not know the product identity (active or placebo) until the end of the study

Exclusion Criteria:

* Reports being pregnant, trying to become pregnant, or breastfeeding
* Unable to provide a valid US shipping address and mobile phone number
* Reports current enrollment in another clinical trial
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Unable to read and understand English
* Reports a current and/or recent (up to 3 months ago) major illness and/or surgery that poses a known, significant safety risk.
* Reports a diagnosis of cardiac dysfunction, liver or kidney disease that presents a known contraindication and/or a significant safety risk with any of the study product ingredients.
* NYHA Class III or IV congestive heart failure, atrial fibrillation, uncontrolled arrhythmias, cirrhosis, end-stage liver disease, stage 3b or 4 chronic kidney disease, or kidney failure
* Reports taking medications that have a well-established moderate or severe interaction, posing a substantial safety risk with any of the study product ingredients.
* Anticoagulants, antihypertensives, anxiolytics, antidepressants, chemotherapy, immunotherapy, sedative hypnotics, medications that warn against grapefruit consumption, corticosteroids at doses greater than 5 mg per day, diabetic medications, oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection, antipsychotics, MAOIs, or thyroid products
* Reports current use of the primary ingredient(s) and/or similar product(s) to the active study product(s) that may limit the effects of the study products and/or pose a safety risk to participants
* Reports an allergy to and/or disinterest in any of the possible study product ingredients
* Lack of reliable daily access to the internet

Ages: 37 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 900 (Actual)
Dates: Start 2025-08-26 (Actual); Primary Completion 2026-01-08 (Actual); Study Completion 2026-01-08 (Actual)

PRIMARY OUTCOMES:
Change in menopausal health issues | 13 weeks
  Difference between rates of change over time in menopausal health issues assessed by Radicle General Menopausal Health Issues (Point range: 6 - 68; where higher scores correspond to more severe menopausal health issues)

SECONDARY OUTCOMES:
Change in feelings of anger | 13 weeks
  Difference between rates of change over time in anger score as assessed by PROMIS Anger 5A (scale 5-25; with higher scores corresponding to more severe anger)
Change in feelings of anxiety | 13 weeks
  Difference between rates of change over time in feelings of anxiety score as assessed by PROMIS Anxiety 8A (scale 8-40; with higher scores corresponding to more severe anxiety)
Change in sleep | 13 weeks
  Difference in rates of change over time in sleep score as assessed by PROMIS Sleep Disturbance 8A (scale 8-40; where higher scores correspond to higher levels of sleep disturbance)

OTHER OUTCOMES:
Minimal clinically important difference (MCID) in menopausal health issues | 13 weeks
  Likelihood of experiencing minimal clinically important difference in menopausal health issues score assessed by Radicle General Menopausal Health Issues (Point range: 6 - 68; where higher scores correspond to more severe menopausal health issues)
Minimal clinically important difference (MCID) in feelings of anger | 13 weeks
  Likelihood of experiencing minimal clinically important difference in anger score as assessed by PROMIS Anger 5A (scale 5-25; with higher scores corresponding to more severe anger)
Minimal clinically important difference (MCID) in feelings of anxiety | 13 weeks
  Likelihood of experiencing minimal clinically important difference in feelings of anxiety score as assessed by PROMIS Anxiety 8A (scale 8-40; with higher scores corresponding to more severe anxiety)
Minimal clinically important difference (MCID) in sleep | 13 weeks
  Likelihood of experiencing minimal clinically important difference in sleep score as assessed by PROMIS Sleep Disturbance 8A (scale 8-40; where higher scores correspond to higher levels of sleep disturbance)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hewlings, Principal Investigator — Radicle Science
Locations (1):
- Radicle Science, Inc, Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Related Info — https://www.radiclescience.com